CLINICAL TRIAL: NCT06756607
Title: The ECOG-ACRIN SUPPORT Trial: Multilevel Intervention to Improve Diverse Enrollment in Cancer Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EAQ223; ECOG-ACRIN-EAQ223 (Other: DCP)
Record Dates: First submitted 2024-11-14; First posted 2025-01-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participant will receive usual care
- Intervention (Experimental): Participant will receive intervention and receive the SUPPORT toolkit.
  Interventions: Other: SUPPORT toolkit

INTERVENTIONS:
Other: SUPPORT toolkit — The SUPPORT toolkit comprises of the SUPPORT CT website and interaction with a SUPPORT navigator.
  Arms: Intervention

SUMMARY:
The purpose of this study is to conduct a Hybrid Type 1 cluster-randomized, roll-out effectiveness-implementation trial in NCORP community oncology practice sites (N= 500 Black and Latino cancer patients) to evaluate the effectiveness of the EA SUPPORT intervention combining CT navigators and CT research literacy tools in improving Black and Latino patient referral and accrual to NCI-supported CTs (primary outcomes) and participant and provider awareness and knowledge of CTs (secondary outcomes) while assessing implementation factors. Also, with the CUSP2CT data, Evaluation, and Coordinating Center, conduct final site evaluation and disseminate the SUPPORT intervention to NCORP community oncology sites, research bases, and affiliated trial networks.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a Hybrid Type 1 cluster-randomized, roll-out effectiveness-implementation trial in NCORP community oncology practice sites (N= 500 Black and Latino cancer patients) to evaluate the effectiveness of the EA SUPPORT intervention combining CT navigators and CT research literacy tools in improving Black and Latino patient referral and accrual to NCI-supported CTs (primary outcomes) and participant and provider awareness and knowledge of CTs (secondary outcomes) while assessing implementation factors. Also, with the CUSP2CT data, Evaluation, and Coordinating Center, conduct final site evaluation and disseminate the SUPPORT intervention to NCORP community oncology sites, research bases, and affiliated trial networks.

ELIGIBILITY:
Inclusion Criteria:

Participant must be ≥ 18 years of age. Participant must self-identify as Black and/or Latino. Participant must be an oncology patient at a participating NCORP. Participant must be eligible to participate in an ECOG-ACRIN clinical trial. Participant must have the ability to understand and the willingness to sign a e-consent document.

Participant must be receiving care at a participating NCORP affiliated community oncology site.

Participant must be English or Spanish speaking to be eligible. Participant must have access to a landline, smartphone, computer, or tablet.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Participant Referral | End of 12 months
  Participant referral to any NCI-supported CT assessed at the end of the 12 months of intervention stage, which will be collected from the referral tracking sheet during the intervention

SECONDARY OUTCOMES:
Participant Accrual | End of 12 months
  Participant accrual assessed at the end of the 12 months of intervention stage, as abstracted from the clinical trials management system and corroborated with abstracted medical records and providers' clinical notes

OTHER OUTCOMES:
Provider Referral | 12 months after the intervention
  Change in provider referral behavior assessed at 12 months after the intervention
Provider Perceptions of Clinical Trials | 12 months after the intervention
  Change in provider perceptions of clinical trials assessed at 12 months after the intervention
Exploratory outcome | 12 months after the intervention
  Participant referral by provider assessed at 12 months after the intervention and participant referral by clinic site assessed at 12 months after the intervention
Exploratory outcome | 12 months after the intervention
  CUSP2CT selected common measures of (a) Participant CT Awareness and Knowledge and (b) Provider CT Awareness and Knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Simon, MD, MPH, Study Chair — Eastern Cooperative Oncology Group
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No